CLINICAL TRIAL: NCT06585683
Title: Tuberculosis Case Finding at the Completion of the CoVPN 3008 Clinical Trial: a Substudy to CoVPN 3008
Brief Title: Post-Trial Tuberculosis Case Finding: A Substudy of CoVPN 3008
Acronym: CoVPN3008TB
Status: Completed | Type: Observational
Sponsor: COVID-19 Prevention Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Other Study IDs: CoVPN 3008 TB substudy; UM1AI068614 (NIH)
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis
Keywords: TB
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Confirmed TB: Participants with confirmed TB will start treatment and have a follow-up visit soon after to check their TB symptoms again and collect blood samples. They will also have a second follow-up visit at week 26 to assess their treatment progress and TB status.
  Interventions: Diagnostic Test: Clinical Evaluation at Day 4; Diagnostic Test: Laboratory Evaluation at Day 4; Diagnostic Test: Clinical Evaluation at week 26; Diagnostic Test: Laboratory Evaluation at week 26
- no TB (control): Participants without TB will have a single follow-up visit to reassess TB symptoms and collect blood samples.
  Interventions: Diagnostic Test: Clinical Evaluation at Day 4; Diagnostic Test: Laboratory Evaluation at Day 4

INTERVENTIONS:
Diagnostic Test: Clinical Evaluation at Day 4 — Participants will undergo an abbreviated physical exam, assessment of concomitant medications, and reassessment for signs/symptoms of TB
Diagnostic Test: Laboratory Evaluation at Day 4 — Peripheral blood samples, including serum, PBMC, and whole blood, are collected from participants. A tongue swab is also collected from each participant.
Diagnostic Test: Clinical Evaluation at week 26 — Participants will undergo another complete physical exam and have their medical (including TB) history, potential TB signs/symptoms, and concomitant medications reassessed. Chest radiography will be obtained for all participants. An assessment of TB outcomes will also be performed.
  Groups: Confirmed TB
Diagnostic Test: Laboratory Evaluation at week 26 — Peripheral blood samples, including serum, PBMC, and whole blood, will be collected. Participants not previously identified as living with HIV will undergo HIV diagnostic testing, while participants living with HIV will have their HIV viral load and CD4+ T-cell count measured.
  Groups: Confirmed TB

SUMMARY:
This substudy aims to identify cases of tuberculosis after the CoVPN 3008 clinical trial is completed.

DETAILED DESCRIPTION:
This observational substudy will involve participants from the CoVPN 3008 trial, regardless of their HIV status, to study tuberculosis (TB). At the start, all participants will be screened for TB, even if they have no symptoms. They will receive chest x-rays and provide sputum samples for TB testing using Xpert Ultra, smear microscopy, and culture.

The study has two main groups. Group 1 includes participants with confirmed TB, and Group 2 includes participants without TB who will act as controls.

Participants with confirmed TB will start treatment and have a first follow-up visit on Day 4 to reassess TB symptoms and collect blood samples. A second follow-up visit will take place at week 26 to evaluate their treatment progress, clinical outcomes, and TB status, ensuring they receive the necessary care.

Participants without TB will have a single follow-up visit on Day 4 to reassess TB symptoms and collect blood samples. The study aims to identify potential biomarkers of TB by analyzing blood samples from both cases and controls, focusing on gene expression linked to TB, including hidden (subclinical) TB.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment into the CoVPN 3008 clinical trial.
* Able and willing to complete the informed consent process: Volunteer demonstrates an understanding of this substudy.
* Willingness to discuss TB status, undergo related testing/monitoring labs, and receive referrals for TB care.

Exclusion Criteria:

* Investigator's concern for difficulty with venous access based on clinical history and physical examination.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will involve approximately 6,000 volunteers who previously participated in the parent study, CoVPN 3008. Although volunteers may meet the inclusion/exclusion criteria, certain medical, psychiatric, occupational, or other conditions could complicate the evaluation of safety and/or immunogenicity, making some individuals unsuitable for enrollment or retention in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 5694 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with TB | Measured at Day 1, Day 4 and week 26
  The 95% confidence interval on the proportion of participants with TB will be estimated using the "score" method
Association parameters of each demographic variable with confirmed TB. | Measured at Day 1, Day 4 and week 26
  Proportions and 95% CIs will be estimated using the score method. A multivariate analysis will also be conducted using generalized linear regression models with TB as the outcome.
Proportion of participants with confirmed TB at the six-month follow visit out of the total number of participants that are screened at the six-month visit and who had confirmed TB at their enrollment visit. | Measured at Day 1, Day 4 and week 26
  Proportion and 95% CI will be estimated using the score method.
Peripheral blood biomarkers associated with diagnosis of TB, including subclinical TB. | Measured at Day 1, Day 4 and week 26
  TB risk scores will be computed from RNA sequencing data generated from each participant's baseline whole-blood sample (Tempus tube) provided upon enrollment into CoVPN 3008. Association of each score with confirmed TB will be assessed using cross-validated ROC curve analysis with area under curve (AUC) 95% CI estimated using the Delong method.

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Garrett, Study Chair — eThekwini CRS / Centre for the AIDS Programme of Research in South Africa (CAPRISA); Philip Kotze, Study Chair — Qhakaza Mbokodo Research Clinic; Sufia Dadabhai, Study Chair — Blantyre CRS / Johns Hopkins Research Project; Nyaradzo Mgodi, Study Chair — University of Zimbabwe Clinical Trials Research Centre
Locations (41):
- Gaborone CRS, Gaborone, Botswana
- Eswatini Prevention Center CRS, Mbabane, Eswatini
- Kenya (3):
  - Moi University Clinical Research Centre, Eldoret
  - Kisumu Crs, Kisumu
  - Kombewa Clinical Research Center, Kisumu
- Malawi (2):
  - Blantyre CRS, Blantyre
  - Malawi CRS, Lilongwe
- South Africa (26):
  - Synergy Biomed Research Institute, East London, Eastern Cape
  - Nelson Mandela Academic Research Unit CRS, Mthatha, Eastern Cape
  - PHOENIX Pharma (Pty) Ltd, Port Elizabeth, Eastern Cape
  - Josha Resarch CRS, Bloemfontein, Free State
  - MeCRU CRS, Ga-Rankuwa, Gauteng
  - Clinical HIV Research Unit (CHRU)/ Helen Joseph CRS, Johannesburg, Gauteng
  - Newtown Clinical Research, Johannesburg, Gauteng
  - Soweto - Bara CRS, Johannesburg, Gauteng
  - Wits RHI Ward 21 CRS, Johannesburg, Gauteng
  - Tembisa Clinic 4 CoVPN CRS, Tembisa, Gauteng
  - CAPRISA eThekwini CRS, Durban, KwaZulu-Natal
  - Tongaat CRS, Durban, KwaZulu-Natal
  - Vulindlela CRS, Durban, KwaZulu-Natal
  - Isipingo CRS, Isipingo, KwaZulu-Natal
  - Qhakaza Mbokodo Research Clinic CRS, Ladysmith, KwaZulu-Natal
  - Aurum Institute Klerksdorp CRS, Klerksdorp, North West
  - Rustenburg CRS, Rustenburg, North West
  - Emavundleni CRS, Cape Town, Western Cape
  - FAM-CRU (Family Clinical Research Unit), Cape Town, Western Cape
  - Groote Schuur HIV CRS, Cape Town, Western Cape
  - Masiphumelele Clinical Research Site (MASI) CRS, Cape Town, Western Cape
  - TASK Central, Cape Town, Western Cape
  - Univeristy of Cape Town Lung CRS Institute, Cape Town, Western Cape
  - TASK Eden, George, Western Cape
  - Kliptown Soweto CRS, Johannesburg
  - PHRU Matlosana CRS, Klerksdorp
- Uganda (4):
  - UVRI-IAVI HIV Vaccine Program LTD. CRS, Entebbe
  - Baylor-Uganda CRS, Kampala
  - Joint Clinical Research Centre, Kampala
  - MU-JHU Research Collaboration CRS, Kampala
- Zambia (4):
  - Cfhrz Crs, Lusaka
  - Matero Reference Clinic CRS, Lusaka
  - UNC Global Projects / Kamwala District Health Centre, Lusaka
  - Zambia Emory HIV Research Project - Ndola CoVPN CRS, Ndola